CLINICAL TRIAL: NCT04095520
Title: Non-Carious Cervical Lesions Restored With Different Etching Methods and New Injectable Composite: One Year Clinical Follow-Up
Brief Title: 12 Months Clinical Follow-up of Non-Carious Cervical Lesions Restored With New Injectable Composite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Alperen Degirmenci, Assistant Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15/ 06.08.2019
Record Dates: First submitted 2019-09-11; First posted 2019-09-19 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Dental Erosion
MeSH Terms: conditions — Tooth Erosion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paste Type Traditional Composite-GC G Aenial Anterior (Active Comparator): Non-carious cervical lesions with shallow depth of less than 3 mm will be restored with microhybrid composite
  Interventions: Procedure: Laser Etching; Procedure: Phosphoric acid etching
- Injectable Composite- GC G Aenial Universal Injectable (Experimental): Non-carious cervical lesions with shallow depth of less than 3 mm will be restored with injectable form composite
  Interventions: Procedure: Laser Etching; Procedure: Phosphoric acid etching

INTERVENTIONS:
Procedure: Laser Etching — Before the restorations, cavities will be etched Er:Cr YSGG laser with 4W output power, water pressure 95% and air pressure 60% with MGG6 tip with the spot size of 600 µm will be used.
Procedure: Phosphoric acid etching — Before the restorations, cavities will be etched with %37 phosphoric acid for 15 seconds.

SUMMARY:
Non-carious cervical lesions are defined as loss of pathological material not associated with caries in the enamel-cement junction of the tooth. The etiology of these lesions has been defined as brush abrasion, acid-induced erosion and abstraction due to microstructure losses due to stress concentration in a particular region of the tooth. These lesions should be restored using minimally invasive techniques. The necessity of restorative treatment is directly related to the size of the lesion, sensitivity and aesthetic requirements. However, restorative procedures are often challenging because the cavity preparation does not provide adequate retention, and often the cervical end margin is positioned under the gingiva. This leads to contamination of the operation site with blood, saliva and gingival fluid.

Several restorative options have been proposed for the treatment of cervical caries-free lesions. However, due to their high aesthetic properties, improved adhesive capacity and mechanical properties, composites have been accepted as the most suitable choice. Clinical studies have demonstrated that marginal adaptation, marginal discoloration, and roughening methods for retention are the most important factors in the clinical performances of composite restorations in cervical lesions. Therefore, injectable composites with wettability and better adaptability to cavity margins have been introduced. However, the low filler contents of fluid composites and their weak mechanical properties compared to conventional composites have led researchers to doubt their use in caries-free cervical lesions. As a result of the developed material technology, injectable composites with high filler which have reduced polymerization shrinkage have been developed with simplified filler procedure. However, investigators have not encountered any studies investigating which etching technique this material will exhibit better clinical performance and comparing it with traditional pasty composites. The aim of this study is to evaluate the clinical performance of traditional paste type and injectable composites which will be made by using two different etching techniques.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cervical lesions in the mouth with multiples of 4 and 4,

  * Patients over 18 years of age and in permanent dentition,
  * Patients who do not have a pulpal or endodontic lesion on their teeth to be treated,
  * Patients without sensitivity to percussion in the teeth to be treated.

Exclusion Criteria:

Patients with any systemic disease,

* Pregnant or suspected pregnancy and also breastfeeding patients,
* Patients who are allergic to any dental material,
* Patients with any periodontal disease,
* Patients with poor oral hygiene,
* In cases where the teeth are exposed to excessive load due to excessive rupture,
* Cervical caries lesions,
* Patients who continue orthodontic treatment,
* Desensitizing agents or fluoride treatment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Evaluation the Changes of Surface Luster | 1st day, 1st week,6th month, 1st year
  Surface luster of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Retention | 1st day, 1st week,6th month, 1st year
  Fractures and retention of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Surface Staining | 1st day, 1st week,6th month, 1st year
  Surface staining of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Color Stability and Translucency | 1st day, 1st week, 6th month, 1st year
  Color Stability and translucency of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Anatomic Form | 1st day, 1st week, 6th month, 1st year
  Anatomic form of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Marginal Adaptation | 1st day, 1st week, 6th month, 1st year
  Marginal adaptation of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Wear | 1st day, 1st week, 6th month, 1st year
  Wear of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Patients View | 1st day, 1st week, 6th month, 1st year
  Patients view of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Postoperative (hyper-)sensitivity and tooth vitality | 1st day, 1st week, 6th month, 1st year
  Postoperative (hyper-)sensitivity and tooth vitality of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Recurrence of Caries, Erosion, Abfraction | 1st day, 1st week, 6th month, 1st year
  Recurrence of Caries, Erosion, Abfraction of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Tooth integrity | 1st day, 1st week, 6th month, 1st year
  Tooth integrity of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.
Evaluation the Changes of Periodontal response | 1st day, 1st week, 6th month, 1st year
  Periodontal response of the restorations will be evaluated and scored according to the FDI Direct Restorations Clinical Criteria Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yuzuncu Yil University, Faculty of Dentistry, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Celik EU, Tunac AT, Yilmaz F. A Randomized, Controlled, Split-mouth Trial Evaluating the Clinical Performance of High-viscosity Glass-ionomer Restorations in Noncarious Cervical Lesions: Two-year Results. J Adhes Dent. 2018;20(4):299-305. doi: 10.3290/j.jad.a40985. PMID 30206572
- [Result] Celik EU, Tunac AT, Yilmaz F. Three-year clinical evaluation of high-viscosity glass ionomer restorations in non-carious cervical lesions: a randomised controlled split-mouth clinical trial. Clin Oral Investig. 2019 Mar;23(3):1473-1480. doi: 10.1007/s00784-018-2575-y. Epub 2018 Aug 17. PMID 30120605